CLINICAL TRIAL: NCT01909245
Title: Islet Transplantation Using a T-Cell Depleting Immunosuppression Induction Regimen
Brief Title: Islet Cell Transplant for Type 1 Diabetes
Acronym: TCD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12446
Record Dates: First submitted 2013-07-22; First posted 2013-07-26 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islet cells; hypoglycemia; hypoglycemia unawareness; islet after kidney transplantation; islet transplant; insulin independence; insulin dependence; labile diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Islets of Langerhans Transplantation; Immunosuppressive Agents; gastrin 17

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm Study (Experimental): Allogenic Human Islet Cell Transplant with immunosuppression
  Interventions: Biological: Allogenic Human Islet Cells; Drug: Immunosuppressive Agents; Drug: Gastrin 17

INTERVENTIONS:
Biological: Allogenic Human Islet Cells — Intraportal (into the liver) infusion of islet cells, with a maximum of three islet transplants.
  Other Names: Islet transplant, islet transplantation
Drug: Immunosuppressive Agents — Anti-rejection medications (to prevent the body from rejecting the islet cells) and other medications to guard against infection and support participant health and/or the health of the transplanted islets.
Drug: Gastrin 17 — Gastrin-17 (or GAST-17) - a gut hormone injected under the skin for 30 days (optional treatment for islet dysfunction).
  Other Names: GAST-17

SUMMARY:
City of Hope National Medical Center, located in Duarte, CA, is hosting a clinical study on islet cell transplantation, an experimental procedure being evaluated as a treatment for patients with type 1 diabetes. Islet cell transplantation involves taking insulin-producing cells from organ donors and transplanting them into the liver of a patient with diabetes. Once transplanted, the islets produce insulin, which can improve blood sugar control and eliminate the need to inject insulin or use an insulin pump.

Anti-thymocyte globulin (ATG) and alemtuzumab (Campath) are anti-rejection medications that work by decreasing a patient's T-cells. T-cells are special white blood cells that recognize and destroy unwanted things like infections but can also attack transplanted cells and organs. Reducing the number of T-cells at the time of transplant may protect islets and improve long-term transplant success. In previous research studies, islet transplantation has been successful in reducing low blood sugar episodes, improving overall blood sugar control, and in some cases, allowing patients with type 1 diabetes to stop taking insulin.

The purpose of this study is to determine if islet cell transplantation using ATG or alemtuzumab, along with additional medications to prevent the body from rejecting the transplanted cells, is a safe and effective treatment for type 1 diabetes. Study participants may receive up to three islet transplants and will be followed for five years to monitor blood sugar control, islet transplant function, and changes in quality of life.

ELIGIBILITY:
Three different categories of patients with Type 1 Diabetes will be considered for study participation:

* Naïve islet transplant alone (nITA) candidates: T1D patients complicated by frequent/severe hypoglycemia, hypoglycemia unawareness, AND/OR otherwise unstable blood glucose control who have not received a previous transplant (except for a failed pancreas more than 6 months prior to screening)
* Repeat transplant (RT) candidates: T1D patients who have received two or fewer previous islet transplants > 1 month prior to screening, but continue to require exogenous insulin treatment or have an HbA1c > 6.5%
* Islet after kidney transplant (IAK) candidates: T1D patients with a history of successful renal transplant > 3 months prior to screening

Inclusion criteria for all candidates:

1. Age 18-68 years
2. Type 1 diabetes mellitus for at least 5 years
3. Ability and willingness to comply with post-transplant regimen, including taking anti-rejection medications, use of reliable contraception, frequent clinic visits, lab tests, careful recording of blood glucose values, insulin doses and medications, and completing detailed follow-up studies

   Additional Inclusion Criteria nITA Candidates Only
4. Unstable blood sugar control characterized by:

   Frequent hypoglycemia (blood glucose ≤ 54 mg/dl more than once per week) -AND/OR- Hypoglycemia unawareness (Clarke score of 4 or more) -AND/OR- One or more severe hypoglycemic episodes in 12 months preceding enrollment. -AND/OR- Erratic blood glucose levels that interfere with daily activities -AND/OR- One or more hospital visits for diabetic ketoacidosis in the 12 months preceding enrollment

   Additional Inclusion Criteria for RT Candidates Only
5. One or two or previous islet transplants > 1 month prior to screening with continuing insulin requirements and/or HbA1c > 6.5%

   Additional Inclusion Criteria for IAK Candidates Only
6. Successful kidney transplant > 3 months prior to screening
7. Stable maintenance immunosuppression consisting of tacrolimus alone or in conjunction with sirolimus, mycophenolate mofetil, myfortic or azathoprine; or cyclosporine in conjunction with sirolimus, mycophenolate mofetil, or myfortic +/- ≤ 10 mg/day corticosteroids
8. No history of acute rejection related to kidney graft in last 12 months and low risk of rejection
9. Under continuing care of physician for kidney graft, who has provided letter in support of candidate's consideration for study participation

Exclusion Criteria:

1. Body Mass Index (BMI) > 33
2. Insulin requirements > 1.2 units/kg/day
3. Known sensitization to both rATG -and- alemtuzumab
4. Significant kidney dysfunction
5. Significant liver/gall bladder disease
6. Significant cardiovascular disease
7. Active proliferative retinopathy
8. High blood pressure despite appropriate treatment
9. High cholesterol/triglycerides despite appropriate treatment
10. Anemia or other blood disorders that require medical treatment
11. WBC <3,000/ul
12. Increased risk of bleeding, other chronic hemostasis disorders, or treatment with chronic anticoagulant therapy
13. Recent unresolved acute infection (except for mild skin infection or nail fungal infection), or chronic infection
14. Epstein-Barr Virus (EBV) IgG negative
15. Any history of malignancy, except for completely resected squamous or basal cell carcinoma of the skin or in situ cancer of the cervix
16. Recent history of non-adherence to medical treatment, or inability to demonstrate capacity to comply with strict blood glycemic control and insulin therapy
17. Psychiatric illness that is untreated, or likely to interfere significantly with study compliance despite treatment
18. Previous organ/tissue transplant, except as noted above
19. Administration of live attenuated vaccines within 2 months of enrollment
20. Presence of a chronic disease that must be chronically treated with a contraindicated agent
21. Use of investigational agents within four weeks of enrollment
22. Active alcohol or substance abuse, including cigarette smoking
23. Pregnant women, women intending future pregnancy, women of reproductive potential who are unable or unwilling to follow effective contraceptive measures prior to study entry and for as long as they are on immunosuppression medication, and women presently breast feeding are excluded
24. Individuals without health insurance
25. History of gastric bypass
26. Any medical condition that in the opinion of the investigator will interfere with safe participation in the trial

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who are insulin independent, hypoglycemia free, AND with hemoglobin A1c < or = 6.5% at 1 year post-transplant | 1 year post-transplant
Proportion of subjects who are insulin independent, hypoglycemia free, AND with hemoglobin A1c < or = 6.5% at 2 years post-transplant | 2 years post-transplant
Proportion of subjects who are insulin independent, hypoglycemia free, AND with hemoglobin A1c < or = 6.5% at 5 years post-transplant | 5 years post-transplant

SECONDARY OUTCOMES:
Proportion of subjects who are free of severe hypoglycemic episodes AND have a hemoglobin A1c < or = 7.0% | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant

OTHER OUTCOMES:
Proportion of subjects experiencing reduction/elimination of hypoglycemic episodes | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Duration of insulin independence | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Proportion of subjects who maintain a positive c-peptide secretion response to glucose/glucagon stimulation | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Change in average daily insulin use compared to baseline | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Decline in insulin intake/100,000 IEQ infused | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Insulin secretion during Intravenous Glucose Tolerance Test (IVGTT), IVGTT+arginine stimulation (IVGTT+AST), Maximum Stimulated Insulin Secretion test (MSIS), and/or Mixed Meal Tolerance Test (MMTT) | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Rate of alloimmune rejection | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Rate of autoimmune reactivation | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence and severity of adverse events related to islet transplant procedure | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence and severity of adverse events related to immunosuppression | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence of change in immunosuppression drug regimen | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence of immune sensitization defined by presence of anti-HLA antibodies post-transplant that were absent pre-transplant | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence of discontinuation of immunosuppression | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Improvement in glucose time within range during continuous glucose monitoring | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Improvement in Personal Glycemic State (PGS) score calculated from continuous glucose monitoring | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant
Incidence of Gastrin-17 use for treatment of islet graft dysfunction AND incidence of change or early discontinuation of Gastrin-17 treatment | +75 days, +6 months, +12 months, and +2, +3, +4 and +5 years post islet transplant

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Result] Aslamy A, Oh E, Ahn M, Moin ASM, Chang M, Duncan M, Hacker-Stratton J, El-Shahawy M, Kandeel F, DiMeglio LA, Thurmond DC. Exocytosis Protein DOC2B as a Biomarker of Type 1 Diabetes. J Clin Endocrinol Metab. 2018 May 1;103(5):1966-1976. doi: 10.1210/jc.2017-02492. PMID 29506054
- See also: City of Hope Islet Cell Transplantation Program — http://www.cityofhope.org/islets